CLINICAL TRIAL: NCT03234179
Title: A Prognosis and Predicting Genetic Study of Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201705110RIND
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Lung Cancer; Genetic Predisposition to Disease
Keywords: Non small cell lung cancer; Genetic study
MeSH Terms: conditions — Lung Neoplasms; Genetic Predisposition to Disease; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples are stored at the lab of NTUH hospital with protected of security. The information of the study subjects will be reached only by investigator of this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is a leading cause of cancer mortality among adults worldwide. The incidence rates of lung cancer among never smoking females in some parts of East Asia are among the highest in the world. The adenocarcinoma of lung being the most frequently identified histological type is more weakly associated with smoking, and often occurs in females and never-smokers. Although family history of lung cancer has been associated with histological subtypes, the inherited susceptibility factors that affect specific histology are unknown.

Genetic factors that determine individual predisposition to lung cancer have been identified via genome-wide association studies. These known common loci, however, explain only a small fraction of the familial risk of lung cancer. The hypothesis of this study is that there are genetic factors that confer inherited susceptibility among patients with primary non-small-cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
To delineate the genetic etiology underlying NSCLC, this study proposes to employ a family-based linkage analysis, together with rich data generated from NGS, to search for disease susceptibility locus for the patients with strong family history of primary NSCLC. By using family pedigrees, linkage analysis will be able to find co-segregation of alleles through multiple generations at a genetic susceptibility locus and a known genetic marker, and then the highly penetrate gene loci may be detected by our study. These gene loci will be a good genetic predictor of NSCLC which should be a great advantage in treatment, prevention and screening of NSCLC in the future.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's family (within third-degree relatives) has at least one diagnosed of primary non-small cell lung cancer.
2. The patient was diagnosed of primary non-small cell lung cancer at the age < 45 years old.

Exclusion Criteria:

1. Patients without the diagnosis of primary non-small cell lung cancer.
2. Patients who are combined with other malignancy and ongoing chemotherapy / radiation therapy.
3. Patients combined with coagulopathy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of primary non small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2037-08-01 (Estimated)

PRIMARY OUTCOMES:
Genetic information of lung cancer patients | One week after the study subjects sign the permit of informed consents
  Collect study subjects' blood sample and analysis with Genome-wide SNP genotyping

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shing Chen, PhD, Study Director — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD to other researchers.